CLINICAL TRIAL: NCT03418987
Title: The Vertebral Vector in a Horizontal Plane. A Simple Way to See in 3D.
Status: Completed | Type: Observational
Sponsor: Tamas Illes (Other)
Responsible Party: Sponsor-Investigator, Tamas Illes, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB - 3D spine
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Scoliosis
Keywords: 3D imaging; vertebral vector; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Deformities of the spinal column: Patients with adolescent idiopathic scoliosis or adult degenerative scoliosis, treated or untreated.
  Interventions: Other: Medical File data analysis

INTERVENTIONS:
Other: Medical File data analysis — Analysis of the 2D/3D spine images (performed with the sterEOS software and the MATLAB software)

SUMMARY:
The diagnosis and classification of scoliosis are almost exclusively based on frontal and lateral radiographs. Current classifications of adolescent or adult idiopathic degenerative scoliosis are based only on the 2D approach. The classifications consider only the lateral deviation and the sagittal alignment and completely ignore all the changes (the axial vertebral rotation and the lateral translation etc ...) in the horizontal plane.

The demand for an accurate assessment of the vertebral rotation in scoliosis is not new. Biplane x-ray images provide insufficient quantitative or qualitative information on the anatomical landmarks needed to determine axial rotation. Several measurement methods have been published, all of which are based on the evaluation of the relative positions of various posterior vertebral elements. The Perdriolle torsiometer is currently the most accepted method in clinical practice, but its reproducibility is very limited and can not be quantified accurately.The horizontal plane deviations are more accurately evaluated by the CT scan, but the systematic use of this method is limited because of its relatively high cost and excessive radiation dose. Expert opinion is also divided on the veracity and reproducibility of CT scan for such measurements.

Given the absence of a definitive and reproducible measurement method for 3D characterization of the vertebral columnar deformities, the investigators introduced the concept and system of vertebral vectors.The vertebral vector technique is currently the only technique in the world that allows the visualization of vertebral column deformities by analyzing each vertebral body and defining characteristic mathematical and geometric parameters that uniquely characterize each vertebrae. A new digital radioimaging technique based on a low dose X-ray detection technology simultaneously creates frontal and lateral whole body radiographic images captured in a standing position, which is the basis of visualization of the vertebral vector.

To examine the two phenotypes of scoliosis, it is necessary to collect the radiological data specific to the disease. After generating the vertebral vectors and obtaining the three-dimensional coordinates, an analysis and an exact mathematical description will be performed. The projections of the curves in the three planes will also be analyzed, with particular attention to the projections in the horizontal planes. Based on the mathematical models and the axial projection of the curves, a new three-dimensional classification can be imagined for the first time not only for adolescent scoliosis, but also for adult degenerative scoliosis.

The main objective of this study is to develop new evidence-based treatments based on the unambiguous understanding of 3D features of vertebral columnar deformities.

ELIGIBILITY:
Inclusion Criteria:

Patients with adolescent idiopathic scoliosis or adult degenerative scoliosis, treated or untreated, radiographed with the EOS system

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with adolescent idiopathic scoliosis or adult degenerative scoliosis, treated or untreated, radiographed with the EOS system
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
x coordinate of the centroid pedicle | 5 years
  Precise spatial localisation of the centroid pedicle, computed with the sterEOS and MATLAB softwares.
y coordinate of the centroid pedicle | 5 years
  Precise spatial localisation of the centroid pedicle, computed with the sterEOS and MATLAB softwares.
z coordinate of the centroid pedicle | 5 years
  Precise spatial localisation of the centroid pedicle, computed with the sterEOS and MATLAB softwares.
Coordinate of the 'A' point of the vector | 5 years
  Spatial coordinate of the initial point of the vector, computed with the sterEOS and MATLAB softwares.
Coordinate of the 'B' point of the vector | 5 years
  Spatial coordinate of the terminal point of the vector, computed with the sterEOS and MATLAB softwares.

CONTACTS AND LOCATIONS:
Overall Officials: Tamas ILLES, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No